CLINICAL TRIAL: NCT03669042
Title: Post-market, Prospective Evaluation of PHOTO-oxidized Decellularized Bovine Pericardium Used as a Patch in Vascular Repair and Reconstruction Surgery
Brief Title: Post-market, Prospective Evaluation of PHOTO-oxidized Bovine Pericardium in Vascular Surgery
Acronym: PHOTO-V
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artivion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHF1801.000-M
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Vascular Diseases; Peripheral Arterial Disease; Hemodialysis Access Failure (Disorder); Carotid Artery Diseases; Abdominal Aortic Aneurism
MeSH Terms: conditions — Vascular Diseases; Peripheral Arterial Disease; Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): All patients will undergo a vascular repair or reconstruction surgery, which requires the use of PhotoFix. The surgical procedures will vary by patient and by underlying etiology. Therefore, PhotoFix implant sites will also vary. In all cases, PhotoFix will be implanted per the Instructions for Use (IFU).
  Interventions: Device: PhotoFix

INTERVENTIONS:
Device: PhotoFix — PhotoFix Patch Implantation

SUMMARY:
The objective of this post-market clinical follow-up study is to evaluate the clinical outcomes of patients receiving PhotoFix as a patch within a vascular repair or reconstruction procedure.

DETAILED DESCRIPTION:
PhotoFix is prepared from bovine pericardium, which is stabilized using a dye-mediated photo-oxidation process and sterilized using aseptic processing techniques. The primary endpoint for patients with carotid artery stenosis (CAS) undergoing carotid endarterectomies (CEA) will be rate of ipsilateral central neurologic events; the primary endpoint for all other vascular procedures will be primary patency. The secondary endpoints include all-cause reoperation rate, device-related reoperation rate, explant rate, restenosis rate, secondary patency (hemodialysis access repair (HAR) only) and survival. A goal of 100 patients will be enrolled at approximately 10 sites. The enrollment period will span a minimum of 8 months from Institutional Review Board (IRB) approval and site activation. Candidates for this study are adults who require vascular repair or reconstruction surgery that necessitates the use of a patch. Patients will be consented pre-operatively and enrolled patients will be followed for approximately 6 months after PhotoFix surgery. Data will be collected at 5 time points: baseline (pre-operatively), intra-operatively, 1 month post-operatively, 3 months post-operatively, and 6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing a vascular procedure which falls within the indications for use and requires the use of PhotoFix Decellularized Bovine Pericardium
* Patient's surgery is anticipated to occur within 60 days of consent
* Patient is ≥18 years old
* Patient is willing and able to comply with the protocol and follow up period
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* Patient's procedure is a revision of a prior arteriotomy or venotomy
* Patient's procedure requires multiple vascular patches in anatomically distinct regions or other prosthetics (e.g. stents)
* Patient has a medical history of abnormal coagulopathy, bleeding, or thromboembolic disease
* Patient has a medical history of severe immunodeficiency disease
* Patient has a medical history of cancer
* Patient has severe visceral disease in heart or active liver disease or icterus
* Patient has a history of cerebrovascular accident (completed stroke) within 3 months of planned surgery
* Patient has a history of atrial fibrillation and requires a patch for carotid endarterectomy repair
* Patient has an active or potential infection at the surgical site
* Patient has used or plans to use immunomodulatory drugs for ≥ 6 months
* Patient has a sensitivity to products of bovine origin
* Patient is currently enrolled in another study
* Patient has a life expectancy of less than 12 months
* Patient is pregnant or breastfeeding or planning on becoming pregnant or unwilling to use medically acceptable methods of birth control
* Patient's procedure is emergent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J. Morrissey, MD, Principal Investigator — Columbia University
Locations (9):
- United States (9):
  - University of Arizona, Tucson, Arizona
  - Iowa Heart Center, Des Moines, Iowa
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Nebraska, Omaha, Nebraska
  - Columbia University, New York, New York
  - Jobst Vascular Institute, Toledo, Ohio
  - Baylor Scott & White, Temple, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Enrolled Patients
Arm/Group | Treatment
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 85
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Central Neurologic Events
Description: For cases of carotid endarterectomy (CEA) only: Percent of patients who experienced at least one of the central neurologic events of interest (transient ischemic attack, amaurosis fugax, stroke, carotid occlusion).
Time Frame: Up to 6 months, post-op
Measure: Count of Participants; unit: Participants
Groups:
- Carotid Artery Stenosis: Indication for surgery was carotid artery stenosis
Arm/Group | Carotid Artery Stenosis
Number analyzed (Participants) | 78
Participants | 2

2. Primary Outcome: Primary Patency
Description: For all other procedures (non-CEAs): Loss of patency includes loss of previously palpable pulses, presentation of recurrent symptoms, a drop in ABI>0.15 in the case of lower limb artery repair, Doppler ultrasound findings of occlusion, angiography of the affected vessel or a combination of these. Loss of patency will also be considered if an intervention to restore or maintain patency is documented.
Time Frame: Up to 6 months, post-op
Measure: Number; unit: participants with primary patency
Groups:
- Peripheral Arterial Disease: Indication for surgery was peripheral arterial disease.
Arm/Group | Peripheral Arterial Disease
Number analyzed (Participants) | 16
participants with primary patency | 16

3. Secondary Outcome: Overall Survival
Description: Percent of patients surviving
Time Frame: Up to 6 months, post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 94
Participants | 94

4. Secondary Outcome: All-Cause Re-operation Rate
Description: Percent of patients requiring re-operations
Time Frame: Up to 6 months, post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 94
Participants | 1

5. Secondary Outcome: Device-Related Re-operation Rate
Description: Percent of patients requiring unplanned re-operations that are documented as possibly, probably or definitely, device-related.
Time Frame: Up to 6 months, post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 94
Participants | 0

6. Secondary Outcome: Explant Rate
Description: Percent of patients requiring device explants. Explants will include the removal of PhotoFix for any reason after implantation.
Time Frame: Up to 6 months, post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 94
Participants | 0

7. Secondary Outcome: Adverse Event Rate
Description: Percent of patients who experienced at least one adverse event.
Time Frame: Up to 6 months, post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 94
Participants | 28

8. Secondary Outcome: Restenosis Rate
Description: Percent of patients who develop stenosis. Stenosis is considered as the recurrence of abnormal narrowing of an artery or vein after corrective surgery. Categorization of stenosis ≥ 50% will occur if data is available.
Time Frame: Up to 6 months, post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 94
Participants | 4

9. Secondary Outcome: Secondary Patency
Description: For all hemodialysis access repairs only: Time from implantation to the point where the access is abandoned.
Time Frame: Up to 6 months, post-op
Population: No patients were enrolled for hemodialysis access repair.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Last visit for enrolled patients was 6 months.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 12/94
Other Adverse Events (participants affected / at risk) | 21/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=94)
Bleeding event (Surgical and medical procedures) | 2 (2)
cardiac event (Cardiac disorders) | 2 (2)
Infection (Infections and infestations) | 4 (4)
Stroke (Vascular disorders) | 2 (2) — The events reported were in one PAD patient and one CAS patient; both were contralateral (not a primary endpoint).
Thrombosis (Vascular disorders) | 1 (1)
Transient Ischemic Attack (Vascular disorders) | 1 (1)
Other (Surgical and medical procedures) | 5 (8)
Symptomatic Carotid Occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=94)
cardiac event (Cardiac disorders) | 3 (3)
Bleeding event (Surgical and medical procedures) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Inflammation/Edema (Blood and lymphatic system disorders) | 1 (1)
Pain (General disorders) | 5 (5)
Other (General disorders) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT03669042/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT03669042/SAP_001.pdf